CLINICAL TRIAL: NCT02905344
Title: The Effectiveness of Using 3D Printed Anatomically Accurate Models to Educate Patients About Surgery: A Survey
Brief Title: Effectiveness of Using 3D Printed Models to Educate Otolaryngology (Ear, Nose, Nose and Throat (ENT)) Patients About Surgery: A Survey
Status: Completed | Type: Observational
Sponsor: University of Notre Dame (Other)
Responsible Party: Sponsor
Other Study IDs: 14-07-1962
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Pathological Conditions, Anatomical; Deviated Nasal Septum
MeSH Terms: conditions — Pathological Conditions, Anatomical

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Control, no anatomical model used for description
- 2: Anatomical model used for description

SUMMARY:
Within the Ear, Nose, and Throat (ENT) medical space, a relatively small number of patients follow through with elective surgeries to fix ailments like a deviated septum or occluded sinus passage. Patient understanding of their diagnosis and treatment plan is integral to compliance, which ultimately yields improved medical outcomes and better quality of life. Here the investigators report the usage of advanced inkjet 3D printing methods to develop a multimaterial replica of the patient's nasal sinus anatomy, derived from clinical X-ray Computed Tomography (CT) data. The final patient education model was developed over several iterations to optimize material properties, anatomical accuracy and overall display. A two arm, single center, randomized, prospective study was then performed in which 50 ENT surgical candidates (and an associated control group, n = 50) were given an explanation of their anatomy, disease state, and treatment options using the education model as an aid. Each patient was then surveyed for their self-rated understanding of their anatomy, disease, and treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects that are 18 years or older.
* Surgeon must have recommended nasal or sinus surgery
* Not excluded as a surgical candidate

Exclusion Criteria:

* Patients who or not able to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult patients considering sinus surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Question: How did the doctor's visualization help you in your understanding of the surgery? | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Liepert, M.D., Principal Investigator — Notre Dame
Locations (1):
- Michiana ENT Specialty Center, South Bend, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be freely shared upon email request.